CLINICAL TRIAL: NCT02287987
Title: Prospective Randomized Trial Comparing Clamp Versus Clampless Robot Assisted Partial Nephrectomy
Brief Title: CLamp vs Off Clamp Kidney During Partial Nephrectomy
Acronym: CLOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alessandro Antonelli, Dr, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOCKBS 1.1
Record Dates: First submitted 2014-10-10; First posted 2014-11-11 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Nephrectomy; Kidney Neoplasm; Glomerular Filtration Rate
Keywords: Renal function; Off-clamp; Partial nephrectomy; Robotic; Hylar clamping
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clamp (Active Comparator): Laparoscopic robot-assisted partial nephrectomy with clamping the renal pedicle during the resection of the tumor
  Interventions: Procedure: Clamp Robotic partial nephrectomy
- Off clamp (Experimental): Laparoscopic robot-assisted partial nephrectomy without clamping the renal pedicle during the resection of the tumor
  Interventions: Procedure: Clampless Robotic partial nephrectomy

INTERVENTIONS:
Procedure: Clamp Robotic partial nephrectomy — Renal artery clamping during partial nephrectomy
  Arms: Clamp
Procedure: Clampless Robotic partial nephrectomy — Robotic partial nephrectomy without renal artery clamping
  Arms: Off clamp

SUMMARY:
Prospective, randomized trial comparing surgical, functional and oncological outcomes between clamp and clamp-less robot assisted partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* normal coagulation trim
* pre operative Glomerular Filtration Rate (GFR) > 60 ml/min
* healty contralateral kidney
* low (4-6) or intermediate (7-10) RENAL score
* availability of Da Vinci Robotic System

Exclusion Criteria:

* altered coagulation trim
* pre operative Glomerular Filtration Rate (GFR) < 60 ml/min
* anatomic or functional solitary kidney
* RENAL score >10

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) variation | 3-6 months
  difference between pre and post operative Glomerular Filtration Rate (GFR)

SECONDARY OUTCOMES:
Feasibility of clampless robotic partial nephrectomy | Duration of the surgical procedure
  number of cases shifted from clampless to clamping procedure; time of suture of the renal parenchyma; overall operative time.
Morbidity of clampless robotic partial nephrectomy | 90 days
  Estimated blood loss; pre/post operative variation of hemoglobin value; overall complications rate; bleeding complications rate
Oncological safety of clampless robotic partial nephrectomy | 15 days
  positive surgical margins rate

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Antonelli, Doctor, Principal Investigator — Spedali Civili di Brescia
Locations (1):
- Clinical Department of Urology, university Hospital Spedali Civili di Brescia, Brescia, Italy

REFERENCES:
- [Background] Thompson RH, Lane BR, Lohse CM, Leibovich BC, Fergany A, Frank I, Gill IS, Blute ML, Campbell SC. Every minute counts when the renal hilum is clamped during partial nephrectomy. Eur Urol. 2010 Sep;58(3):340-5. doi: 10.1016/j.eururo.2010.05.047. Epub 2010 Jun 9. PMID 20825756
- [Background] Ficarra V, Minervini A, Antonelli A, Bhayani S, Guazzoni G, Longo N, Martorana G, Morgia G, Mottrie A, Porter J, Simeone C, Vittori G, Zattoni F, Carini M. A multicentre matched-pair analysis comparing robot-assisted versus open partial nephrectomy. BJU Int. 2014 Jun;113(6):936-41. doi: 10.1111/bju.12570. Epub 2014 May 22. PMID 24219227
- [Background] Minervini A, Siena G, Antonelli A, Bianchi G, Bocciardi AM, Cosciani Cunico S, Ficarra V, Fiori C, Fusco F, Mari A, Martorana G, Medica M, Mirone V, Morgia G, Porpiglia F, Rocco F, Rovereto B, Schiavina R, Simeone C, Terrone C, Volpe A, Carini M, Serni S; Members of the RECORd Project-LUNA Foundation. Open versus laparoscopic partial nephrectomy for clinical T1a renal masses: a matched-pair comparison of 280 patients with TRIFECTA outcomes (RECORd Project). World J Urol. 2014 Feb;32(1):257-63. doi: 10.1007/s00345-013-1155-7. Epub 2013 Sep 7. PMID 24013181
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Kaczmarek BF, Tanagho YS, Hillyer SP, Mullins JK, Diaz M, Trinh QD, Bhayani SB, Allaf ME, Stifelman MD, Kaouk JH, Rogers CG. Off-clamp robot-assisted partial nephrectomy preserves renal function: a multi-institutional propensity score analysis. Eur Urol. 2013 Dec;64(6):988-93. doi: 10.1016/j.eururo.2012.10.009. Epub 2012 Oct 16. PMID 23122834
- [Background] Kutikov A, Uzzo RG. The R.E.N.A.L. nephrometry score: a comprehensive standardized system for quantitating renal tumor size, location and depth. J Urol. 2009 Sep;182(3):844-53. doi: 10.1016/j.juro.2009.05.035. Epub 2009 Jul 17. PMID 19616235
- [Background] Minervini A, Carini M, Uzzo RG, Campi R, Smaldone MC, Kutikov A. Standardized reporting of resection technique during nephron-sparing surgery: the surface-intermediate-base margin score. Eur Urol. 2014 Nov;66(5):803-5. doi: 10.1016/j.eururo.2014.06.002. Epub 2014 Jun 18. PMID 24954792
- [Derived] Bertolo R, Bove P, Sandri M, Celia A, Cindolo L, Cipriani C, Falsaperla M, Leonardo C, Mari A, Parma P, Veccia A, Veneziano D, Minervini A, Antonelli A; AGILE Group (Italian Group for Advanced Laparoendoscopic Surgery). Randomized Clinical Trial Comparing On-clamp Versus Off-clamp Laparoscopic Partial Nephrectomy for Small Renal Masses (CLOCK II Laparoscopic Study): A Intention-to-treat Analysis of Perioperative Outcomes. Eur Urol Open Sci. 2022 Oct 28;46:75-81. doi: 10.1016/j.euros.2022.10.007. eCollection 2022 Dec. PMID 36506251
- [Derived] Antonelli A, Cindolo L, Sandri M, Bertolo R, Annino F, Carini M, Celia A, D'Orta C, De Concilio B, Furlan M, Giommoni V, Ingrosso M, Mari A, Muto G, Nucciotti R, Porreca A, Primiceri G, Schips L, Sessa F, Simeone C, Veccia A, Minervini A; AGILE Group (Italian Group for Advanced Laparo-Endoscopic Surgery). Safety of on- vs off-clamp robotic partial nephrectomy: per-protocol analysis from the data of the CLOCK randomized trial. World J Urol. 2020 May;38(5):1101-1108. doi: 10.1007/s00345-019-02879-4. Epub 2019 Jul 24. PMID 31342246
- See also: EAU guidelines 2014 — http://www.uroweb.org/guidelines